CLINICAL TRIAL: NCT04951102
Title: An Electronic Shared Decision-Making Application to Improve Asthma Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alan Baptist, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00193830
Record Dates: First submitted 2021-06-04; First posted 2021-07-06 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Asthma
Keywords: Asthma; Shared Decision Making; SDM
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The subjects will be clustered in 2 groups of patients and physicians based on participating health care provider and clinic location. Group A will be the intervention group and Group B will be the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A Patients who receive SDM intervention (Experimental): Group A patients will complete a pre-visit electronic Asthma SDM App. They may also receive educational information regarding asthma, medication management, smoking cessation, COVID-19 and COVID-19 vaccines.
  Interventions: Behavioral: Electronic Asthma Shared Decision-Making App
- Group B Patients who receive standard care (Active Comparator): Group B patients will receive standard care.
  Interventions: Behavioral: Standard Care
- Group A Physicians who receive SDM training and electronic Asthma SDM App data (Experimental): Group A physicians will view an SDM Physician Training Video and receive the patients' reported data from the pre-visit asthma SDM App prior to the patients' visits.
  Interventions: Behavioral: Shared Decision Making Physician Training Video; Behavioral: Electronic Asthma Shared Decision-Making App- Patient Data
- Group B Physicians who provide standard care (Active Comparator): Group B physicians will provide standard care.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Electronic Asthma Shared Decision-Making App — The electronic Asthma SDM App will ask questions related to medicine-related, non-medicine-related, and COVID-19-related concerns about patients' asthma, the patients' personal goals for asthma control and expectation for their upcoming visit, and the patients' preferred level of details and involvement in coming to a decision about their asthma treatment. They may also use the Asthma SDM app to find information about asthma, medication management, COVID-19 and COVID-19 vaccines.
  Arms: Group A Patients who receive SDM intervention
Behavioral: Shared Decision Making Physician Training Video — Training video to educate physicians on Shared Decision-Making and the use of Shared Decision-Making tools.
  Arms: Group A Physicians who receive SDM training and electronic Asthma SDM App data
Behavioral: Electronic Asthma Shared Decision-Making App- Patient Data — Data from the pre-visit electronic Asthma SDM app completed by the patients. Data includes medicine-related, non-medicine-related, and COVID-related concerns about patients' asthma, the patients' personal goals for asthma control and expectation for their upcoming visit, and the patients' preferred level of details and involvement in coming to a decision about their asthma treatment.
  Arms: Group A Physicians who receive SDM training and electronic Asthma SDM App data
Behavioral: Standard Care — Standard Care for asthma.
  Arms: Group B Patients who receive standard care; Group B Physicians who provide standard care

SUMMARY:
This study will increase knowledge about the feasibility and effect on patient satisfaction and clinical outcomes of using an electronic Shared Decision Making (SDM) application (app) for patients with asthma in the allergy/immunology clinic visit setting. SDM is defined as an approach where clinicians and patients share the best available evidence when faced with the task of making decisions, and where patients are supported to consider options and make informed choices.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of persistent asthma
* Have an in-person visit or telehealth encounter at the allergy/clinical immunology clinics participating in this study

Exclusion Criteria:

* Diagnosis of intermittent asthma
* Any other lung disease
* Smoking greater than 20 pack years or current smoking
* Mental impairment such that participation would not be possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Within 1 week of completing asthma shared decision making app worksheet and their asthma clinic visit
  Patient satisfaction as determined by Patient Satisfaction Questionnaire responses. Questions will consist of the SDM-Q-9 (psychometrically validated measures for shared decision-making from the perspectives of patients), questions regarding satisfaction with content covered during the visit, and questions regarding satisfaction with the overall communication between the patient and physician.

SECONDARY OUTCOMES:
Physician satisfaction | Within 1 week of patient visit
  Physician satisfaction as determined by Physician Satisfaction Questionnaire responses. Questions will consist of the SDM-Q-DOC (psychometrically validated measures for shared decision-making from the perspectives of health care providers), questions regarding satisfaction with content covered during the visit, and questions regarding satisfaction with the overall communication between the patient and physician. Physicians will receive a small number of satisfaction questionnaires, randomly assigned after patient visits, no more than one a week.
Change in level of asthma control will be determined | Up to 6 months
  Change in level of asthma control as determined by patient follow up asthma control test questionnaire responses regarding interval changes in asthma control, use of systemic steroids, and urgent care and emergency visits for asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Baptist, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee DL, Hammond JW, Finkel K, Gardner DD, Nelson B, Baptist AP. An Electronic Shared Decision-Making App to Improve Asthma Outcomes: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2023 Oct;11(10):3116-3122.e5. doi: 10.1016/j.jaip.2023.06.016. Epub 2023 Jun 16. PMID 37329951